CLINICAL TRIAL: NCT04295421
Title: Comparison of Adductor Canal Block and IPACK Block With Adductor Canal Block Alone After Total Knee Arthroplasty
Brief Title: IPACK Block After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Collaborators: Institut Kassab d'Orthopédie (Other)
Responsible Party: Principal Investigator, Olfa kaabachi, MD, Professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE-IMKO 101/2019
Record Dates: First submitted 2020-02-24; First posted 2020-03-04 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Knee Arthropathy; Postoperative Pain
Keywords: knee arthoplasty; nerve block; analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Canal adductor block (Active Comparator): ACB was done in the immediate postoperative period under a high-frequency ultrasound guidance in which the adductor canal was identified beneath the sartorius muscle and 20 ml of 0.2% ropivacaine was injected in the canal using a 22-gauge 100-mm short-beveled regional block needle and a catheter was kept for 48H with 4 ml/h ropivacaine 0.2%.
  Interventions: Procedure: adductor canal block
- IPACK block (Experimental): IPACK was realized after spinal anesthesia. Patient was placed in a supine position and knee placed in position of 90° flexion. A low-frequency ultrasound probe was positioned in the popliteal crease, and the needle was inserted from medial aspect of the knee from anteromedial to posterolateral direction in a plane between the popliteal artery and the femur. The tip of the needle was placed 1-2 cm beyond the lateral edge of the artery, and 20 ml of 0.2% ropivacaine was injected for each side.
  A ACB was done postoperatively with 20 ml ropivacaine 0.2% and a catheter was kept for 48H with 4 ml/h saline
  Interventions: Procedure: adductor canal block; Procedure: IPACK block

INTERVENTIONS:
Procedure: adductor canal block — ACB was done in the immediate postoperative period under a high-frequency ultrasound guidance in which the adductor canal was identified beneath the sartorius muscle and 20 ml of 0.2% ropivacaine was injected in the canal using a 22-gauge 100-mm short-beveled regional block needle and a catheter was kept for 48H with 4 ml/h ropivacaine 0.2%.
Procedure: IPACK block — IPACK block was realized after spinal anesthesia with 40 ml 0.2% ropivacaine and at the end of surgery , patients were given ACB with 20 ml 0.2% ropivacaine and continued with 4 ml/H saline for 48H
  Arms: IPACK block

SUMMARY:
Adductor canal block (ACB) is a peripheral nerve blockade technique that provides good pain control in patients undergoing total knee arthroplasty (TKA) which however does not relieve posterior knee pain. The recent technique of an ultrasound-guided local anesthetic infiltration of the interspace between popliteal artery and the capsule of posterior knee (IPACK) has shown promising results in providing significant posterior knee analgesia without affecting the motor nerves. The hypothesis was that the combination of ACB + IPACK will provide better pain relief and improve knee function in the immediate postoperative period compared to ACB alone.

DETAILED DESCRIPTION:
This is a prospective, randomized and double blinded study

All patients received :

* Pregabalin 150 mg preoperatively 12 h before the surgery.
* Single-shot spinal anesthesia with 10 to 12 mg of bupivacaine 0.5% and 2.5ug sufentanil patients were randomly allocated to receive:
* Group 1: IPACK + ACB single shoot
* Group 2: contineous ACB For group 1: IPACK was realized after spinal anesthesia with 40 ml ropivacaine 0.2% All patients received ACB in the immediate postoperative period with 20 ml ropivacaine 0.2%

Post operative analgesia included:

* Paracetamol 1g IV every 6 hours
* Diclofenac sodium (50mg) 1 tablet x 2 per day
* Pregabalin 150 mg given orally once daily for a period of 4 weeks.
* PCA morphine (Patient Controlled Analgesia), as a rescue analgesia,
* Continuous ACB catheter for 48H with :

  4 ml per hour 0.2% ropivacaine in group 2 4 ml per hour saline in group 1

ELIGIBILITY:
Inclusion Criteria:

* primary total knee arthroplasty under spinal anesthesia

Exclusion Criteria:

* Contraindication or refusal to regional anesthesia
* Contraindication to non steroidal anti inflammatory (NSAID's)
* Allergy to opioids
* Allergy to paracetamol
* Creatinine clearance < 30ml/min
* Weight<50 kg or >100kg

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | Day 2
  total Morphine consumption

SECONDARY OUTCOMES:
Pain score at rest | Day 2
  numerical rating scale [0=no pain ; 10=worste pain]
Pain score during mouvment | Day 2 [0=no pain ; 10=worste pain]
  numerical rating scale
Ambulation distance | Day 2
  number of steps walked by the patient
Chronic pain | Month 6
  DN4 score [0=minimum to 10= worste score]
functional status | Month 6
  KOOS PS score [0=minimum to 28= worste score]

CONTACTS AND LOCATIONS:
Overall Officials: khaireddine Raddaoui, MD, Principal Investigator — Tunis El Manar University
Locations (1):
- Institut Kassab D'Orthopedie, Tunis, Tunisia